CLINICAL TRIAL: NCT06308432
Title: Sweat Rate Measurement With a Sensor (Wearable) in Different Climatic Conditions With Road Cyclists.
Acronym: CYSU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Francisco Javier López Román, Principal Investigator, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: UCAMCFE-00036
Record Dates: First submitted 2024-02-15; First posted 2024-03-13 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-01

CONDITIONS: Sweat
Keywords: Cyclist; Performance; Temperature; Humidity
MeSH Terms: interventions — Ultrasonic Waves; Cold Temperature; SLH1 protein, Arabidopsis; Diathermy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 22 degrees, 40% humidity and 50% intensity (Experimental): The room in which the 30-minute test will be performed will be at 22 degrees Celsius and 40% humidity.
  The subject should perform the test at 50% of the power at which he reached his VO2max.
  Interventions: Other: Low intensity; Other: Low temperature; Other: Low Humidity
- 35 degrees, 40% humidity and 50% intensity (Experimental): The room in which the 30-minute test will be performed will be at 35 degrees Celsius and 40% humidity.
  The subject should perform the test at 50% of the power at which he reached his VO2max.
  Interventions: Other: Low intensity; Other: Low Humidity; Other: High temperature
- 35 degrees, 65% humidity and 50% intensity (Experimental): The room in which the 30-minute test will be performed will be at 35 degrees Celsius and 65% humidity.
  The subject should perform the test at 50% of the power at which he reached his VO2max.
  Interventions: Other: Low intensity; Other: High temperature; Other: High humidity
- 22 degrees, 40% humidity and 60% intensity (Experimental): The room in which the 30-minute test will be performed will be at 22 degrees Celsius and 40% humidity.
  The subject should perform the test at 60% of the power at which he reached his VO2max.
  Interventions: Other: Low temperature; Other: Low Humidity; Other: High intensity
- 35 degrees, 40% humidity and 60% intensity (Experimental): The room in which the 30-minute test will be performed will be at 35 degrees Celsius and 40% humidity.
  The subject should perform the test at 60% of the power at which he reached his VO2max.
  Interventions: Other: Low Humidity; Other: High intensity; Other: High temperature
- 35 degrees, 65% humidity and 60% intensity (Experimental): The room in which the 30-minute test will be performed will be at 35 degrees Celsius and 65% humidity.
  The subject should perform the test at 60% of the power at which he reached his VO2max.
  Interventions: Other: High intensity; Other: High temperature; Other: High humidity

INTERVENTIONS:
Other: Low intensity — The subject will perform the 30-minute test at an intensity of 50% of the power at which he/she has reached his/her VO2max.
  Arms: 22 degrees, 40% humidity and 50% intensity; 35 degrees, 40% humidity and 50% intensity; 35 degrees, 65% humidity and 50% intensity
Other: Low temperature — The performance test will be carried out in a room conditioned to a temperature of 22º.
  Arms: 22 degrees, 40% humidity and 50% intensity; 22 degrees, 40% humidity and 60% intensity
Other: Low Humidity — The performance test will be carried out in a room conditioned to 40% humidity.
  Arms: 22 degrees, 40% humidity and 50% intensity; 22 degrees, 40% humidity and 60% intensity; 35 degrees, 40% humidity and 50% intensity; 35 degrees, 40% humidity and 60% intensity
Other: High intensity — The subject will perform the 30-minute test at an intensity of 60% of the power at which he/she has reached his/her VO2max.
  Arms: 22 degrees, 40% humidity and 60% intensity; 35 degrees, 40% humidity and 60% intensity; 35 degrees, 65% humidity and 60% intensity
Other: High temperature — The performance test will be carried out in a room conditioned to a temperature of 35º.
  Arms: 35 degrees, 40% humidity and 50% intensity; 35 degrees, 40% humidity and 60% intensity; 35 degrees, 65% humidity and 50% intensity; 35 degrees, 65% humidity and 60% intensity
Other: High humidity — The performance test will be carried out in a room conditioned to 65% humidity.
  Arms: 35 degrees, 65% humidity and 50% intensity; 35 degrees, 65% humidity and 60% intensity

SUMMARY:
Controlled, double-blind, crossover clinical trial with six parallel arms depending on the combination of temperature and humidity (22º and 40% humidity, 35º 40% humidity and 35º and 65% humidity), with two differents intensity, to investigate and validate the physiological use of a sensor in recreational road cyclists.

DETAILED DESCRIPTION:
Subjects who meet the inclusion criteria will be recruited to participate in the clinical trial and perform the exercise sessions.

The cyclists in the study will have to make 7 visits to the laboratory. At the first visit, their aerobic performance will be evaluated by an incremental test to exhaustion with gas analysis. And in the next 6 visits they will have to perform a sustained intensity exercise with different environmental conditions according to the combination of temperature, humidity and intensity.

ELIGIBILITY:
Inclusion Criteria:

* Male cyclists with more than two years of cycling experience.
* Perform tests without fatigue.
* Road bike training at least twice a week.

Exclusion Criteria:

* Participants with chronic illness.
* Have a long-term injury that prevents you from training in the previous month.
* Inability to understand informed consent.
* Use of diuretics in the month prior to or during the measurement period.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2024-02-19 (Actual); Primary Completion 2024-04-12 (Actual); Study Completion 2024-05-20 (Actual)

PRIMARY OUTCOMES:
Sweat | Change of baseline rate of sweet rate in six occasions (the first day, day 7, day, 14, day 21, day 28, day 35)
  The amount of sweat will be measured by a sensor placed on the back.

SECONDARY OUTCOMES:
Microcapillary Blood | Change of baseline rate of sweet rate in six occasions (the first day, day 7, day, 14, day 21, day 28, day 35)
  By means of a lancet puncture in the thumb of the finger, 70 ml of capillary blood will be extracted.This test provides biochemical variables (ABL90FLEX) with 70 ml of capillary blood.
Heart Rate | Changes of heart rate in six occasions (the first day, day 7, day, 14, day 21, day 28, day 35)
  The heart rate will be evaluated by means of a heart rate strap.
Fatigue | Change of fatigue in six occasions (the first day, day 7, day, 14, day 21, day 28, day 35)
  Rate of perceived exertion using Borg scale. En esta escala 0 representa nada fatigado y el 10 esfuerzo máximo.
Temperature on the forehead | Changes in Temperature on the forehead in six occasions (the first day, day 7, day, 14, day 21, day 28, day 35)
  The temperature will be measured by an infrared thermometer.
Temperature in the ear | Changes in Temperature in the ear in six occasions (the first day, day 7, day, 14, day 21, day 28, day 35)
  The temperature will be measured by ear thermometer.
Sleep efficiency | Changes in the sleep efficiency in six occasions (the first day, day 7, day, 14, day 21, day 28, day 35)
  Measured by accelerometry, with Actigraph wGT3X-BT
Karolinska drowsiness scale | It will be measured the day after in six occasions (the first day, day 7, day, 14, day 21, day 28, day 35)
  Measured by Karolinska test

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of Murcia, Murcia, Spain